CLINICAL TRIAL: NCT04510870
Title: Iron Deficiency as an Ignored Cause of Infertility
Acronym: IDI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dextra Fertility Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FI028.DEX001.2019; 2019-002040-24 (EudraCT Number); KLnro136/2019 (Other: Finnish Medicines Agency FIMEA)
Record Dates: First submitted 2020-08-09; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Iron Deficiency; Infertility
Keywords: low ferritin; infertility; in vitro fertilization (IVF); intracytoplasmic sperm injection (ICSI); assisted reproductive technology (ART)
MeSH Terms: conditions — Iron Deficiencies; Infertility | interventions — ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 1. infusion is ferric carboxymaltose, dosage according to the summary of product characteristics (SmPC)
  2. infusion is NaCl
  Interventions: Drug: Ferric Carboxymaltose Injection; Drug: NaCl infusion
- NaCl infusion group (Experimental): 1. infusion is NaCl
  2. infusion is ferric carboxymaltose, dosage according to the summary of product characteristics (SmPC)
  Interventions: Drug: Ferric Carboxymaltose Injection; Drug: NaCl infusion

INTERVENTIONS:
Drug: Ferric Carboxymaltose Injection — Infusion prior the start of IVF/ICSI cycle. Dosing according to the summary of product characteristics (SmPC) chart. Placebo infusion before frozen embryo transfer if needed.
  Other Names: Ferinject
Drug: NaCl infusion — Placebo infusion prior the start of IVF/ICSI cycle. Ferric Carboxymaltose infusion before frozen embryo transfer if needed. Dosing according to the summary of product characteristics (SmPC) chart.

SUMMARY:
Iron deficiency may play a critical role in human infertility, oocyte quality and may even play a role in endometrial receptivity. By correcting iron deficiency, low ferritin values, in infertile women with intravenous iron supplementation, embryo quality and pregnancy rates may improve.

The main objective is to evaluate the effect of intravenous iron supplementation on embryo quality (number of good quality blastocysts).

Randomized, double blind, parallel group, cross-over study of ferric carboxymaltose compared to placebo (NaCl infusion).

ELIGIBILITY:
Inclusion Criteria:

* Patient's 18 to 42 years and in full consent
* Ferritin ≤ 30 ug/l
* Anti-mullerian hormone (AMH) > 1ug/l
* Planned for IVF/ ICSI treatment
* Diagnosis for treatment: tubal factor, male factor or unexplained infertility (NUD)

Exclusion Criteria:

* Endometriosis
* Poor responder
* Inflammatory bowel disease (IBD), colitis ulcerosa
* Rheumatoid arthritis
* Renal insufficiency
* Cardiac insufficiency
* Body Mass Index (BMI) over 35
* Known hypersensitivity to the active substance, to ferric carboxymaltose or any of its excipients, or to other parental iron products
* Clinical evidence of iron overload or disturbances in the utilization of iron
* use of atosiban or filgrastim during stimulation or embryo transfer

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — evaluates female part in reproduction
Enrollment: 62 (Estimated)
Dates: Start 2020-08-17 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of good quality blastocysts | day 5-7 after oocyte pick up
  good quality blastocyst are defined as blastocyst, which are transferable or may be frozen

SECONDARY OUTCOMES:
blastulation rate | day 5-7 after oocyte pick up
  number of blastocysts /fertilized oocyte
ongoing pregnancy/ pregnancy rate | 10 weeks after oocyte pick up,at oocyte pick up it counted to be 2 weeks of gestation.
  ongoing pregnancy at 12 weeks of gestation/ positive pregnancy test (%)
mature oocyte rate | 1 day after oocyte pick up
  number of mature oocytes / total number of oocytes (%)
fertilization rate | 1 day after oocyte pick up
  number of fertilized oocytes/total number of oocytes (%)
implantation rate | 5 weeks after embryo transfer
  number of attached embryos/ embryo transfer (%)

OTHER OUTCOMES:
endometrial thickness | 1 month after infusion, at the time of embryo transfer
  difference of endometrial thickness in mm compared at the day of infusion and the day of embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Annika Tulenheimo-Silfvast, M.D, Principal Investigator — senior consultant
Locations (1):
- Dextra Fertility Clinic, Helsinki, Finland